CLINICAL TRIAL: NCT07392229
Title: Zanubrutinib, a Second Generation BTK Inhibitor, in Anti-MAG Antibody Neuropathy: a Phase II Italian Multicenter Clinical Trial (MAZINGA)
Brief Title: Zanubritnib and Anti-MAG Neuropathy
Acronym: MAZINGA
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Azienda Ospedaliera di Padova (Other)
Collaborators: ClinOpsHub Srl (CRO) (Unknown)
Responsible Party: Principal Investigator, Dr Andrea Visentin, Principal Investigator, Azienda Ospedaliera di Padova
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MAZ-01
Record Dates: First submitted 2026-01-21; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Anti-MAG IgM-associated Demyelinating Polyneuropathy
MeSH Terms: interventions — zanubrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment arm (Experimental)
  Interventions: Drug: Zanubrutinib Oral Capsule

INTERVENTIONS:
Drug: Zanubrutinib Oral Capsule — ZANUBRUTINIB ORAL CAPSULES or Brukinsa Oral Capsule

SUMMARY:
The MAZINGA study is a multicenter, open-label, single-arm Phase IIA clinical trial designed to evaluate the efficacy, safety, and tolerability of zanubrutinib in patients with IgM anti-myelin-associated glycoprotein (anti-MAG) antibody-associated demyelinating polyneuropathy. Anti-MAG neuropathy is a rare immune-mediated disorder frequently associated with IgM monoclonal gammopathies, including monoclonal gammopathy of undetermined significance (MGUS), Waldenström macroglobulinemia, marginal zone lymphoma, chronic lymphocytic leukemia, and other indolent B-cell lymphoproliferative disorders.

The primary objective of the study is to determine whether 12 months of treatment with zanubrutinib leads to a clinically meaningful neurological improvement, defined as an improvement of at least one point in at least two validated neurological scales. These include reductions in the Overall Neuropathy Limitations Scale (ONLS), INCAT Disability Score, and INCAT Sensory Sum Score (ISS), along with increases in the Medical Research Council (MRC) sum score and the I-RODS functional score.

Secondary objectives include the evaluation of neurophysiological improvement assessed by nerve conduction studies (ENG/EMG), particularly changes in distal motor latency, terminal latency index, and sensory action potential amplitude at 12, 24, and 48 months. Additional secondary endpoints assess hematological efficacy through overall response rate (complete response, very good partial response, or partial response), event-free survival, time to neurological progression, and overall survival. The safety profile of zanubrutinib will be characterized by the incidence, type, and severity of adverse events, serious adverse events, and events of special interest.

Eligible participants are adults (≥18 years) with a confirmed diagnosis of anti-MAG IgM-associated demyelinating polyneuropathy, evidence of a relevant IgM monoclonal gammopathy, elevated anti-MAG antibody titers, and measurable neurological disability. Both treatment-naïve and relapsed/refractory patients are eligible. Key exclusion criteria include prior treatment with BTK inhibitors, aggressive lymphomas, significant axonal damage, uncontrolled comorbidities, active infections, pregnancy, or conditions that could interfere with study participation or safety evaluation.

The planned sample size is approximately 50 patients recruited from nine Italian centers. Statistical analyses will compare neurological outcomes with historical controls, estimate survival endpoints using Kaplan-Meier methods, and explore associations between clinical outcomes and molecular features. This study aims to provide robust prospective evidence on the role of BTK inhibition in anti-MAG neuropathy and to inform future therapeutic strategies for this rare and disabling condition.

ELIGIBILITY:
Inclusion Criteria (MAIN):

* age ≥18 years;
* diagnosis of anti-MAG antibody polyneuropathy;
* neurophysiological (ENG/EMG) evidence of a demyelinating polyneuropathy with evidence of disproportionately prolonged distal motor latency in one or more nerves -excluding the median nerve if related to carpal tunnel syndrome
* IgM monoclonal protein underlying MGUS (based on the WHO definition of clonal lympho- plasmocytes <10%), Waldenstrom macroglobulinemia (based on the WHO definition of clonal lympho-plasmocytes ≥10%), marginal zone lymphoma, chronic lymphocytic leukemia or low- grade lymphoma not otherwise specified;
* presence of anti MAG antibodies (titer ≥ 7.000 BTU);
* neurophysiological (ENG/EMG) evidence of demyelinating polyneuropathy.

Exclusion Criteria (MAIN):

* Previous treatment with BTK inhibitors
* Aggressive non-Hodgkin lymphoma or IgM multiple myeloma
* Evidence of moderate or severe motor nerve axonal damage, defined when occurring diffuse polyneuropathic denervation or a recruitment pattern lower than intermediate in ≥50% of muscles examined, and/or INCAT at lower limbs ≥4.
* ECOG >3
* Use of strong CYP3A inducers within 14 days prior to the first dose of zanubrutinib

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-05-04 (Estimated); Primary Completion 2031-03 (Estimated); Study Completion 2031-03 (Estimated)

PRIMARY OUTCOMES:
The proportion of patients with neurological improvement defined as improvement of at least 1 point after 12 months of zanubrutinib treatment. | 5 years

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2025-12-03): https://cdn.clinicaltrials.gov/large-docs/29/NCT07392229/Prot_000.pdf